CLINICAL TRIAL: NCT06369662
Title: Prognostic and Predictive Values of CD155 in Patients With Acute Myeloid Leukemia
Brief Title: CD155 Expression in Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nehal Adel Rayan Mohamed, Assistant Lecturer, Assiut University
Other Study IDs: SECI-CD155; SECI-IRB-IORG0006563-545 (Other: Scientific Research Unit)
Record Dates: First submitted 2021-07-12; First posted 2024-04-17 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Neoplasms; Hematologic Neoplasms; Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute
Keywords: CD155; AML; Survival
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms; Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Peripheral blood or Bone marrow aspiration specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AML Patients: Adult patients (from 18 - 60 years) diagnosed as AML
  Interventions: Diagnostic Test: Flow cytometric immunophenotyping; Diagnostic Test: Complete blood count; Diagnostic Test: Bone marrow aspiration; Diagnostic Test: Cytogenetic testing; Diagnostic Test: FLT3-ITD using High resolution melting curve (HRM) analysis

INTERVENTIONS:
Diagnostic Test: Flow cytometric immunophenotyping — CD155 expression by flow cytometric immunophenotyping
Diagnostic Test: Complete blood count — Complete blood count with peripheral blood smear examination
Diagnostic Test: Bone marrow aspiration — Bone marrow aspiration at both diagnosis and follow up of patients
Diagnostic Test: Cytogenetic testing — Karyotyping or AML fluorescence in situ hybridization (FISH) panel for diagnosis and risk stratification of AML patients
Diagnostic Test: FLT3-ITD using High resolution melting curve (HRM) analysis — Detection of FLT3-ITD mutation in AML patinets

SUMMARY:
Acute myeloid leukemia (AML) is a heterogeneous hematologic malignancy. It is the most common form of acute leukemia among adults. In the United States, an estimated 19,940 people will be diagnosed with AML in 2020.

CD155 expression was associated with an unfavorable prognosis in solid tumors such as colon cancer, breast cancer, lung adenocarcinoma, pancreatic cancer, melanoma, and glioblastoma, as it correlated with tumor migration, development of metastases, tissue and lymph node invasion, relapse, and poorer survival.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a heterogeneous hematologic malignancy. It is the most common form of acute leukemia among adults. In the United States, an estimated 19,940 people will be diagnosed with AML in 2020.

T-cell exhaustion is a state of decline in T-cell proliferation and function (secretion of cytokines and cytotoxicity). It is defined by the expression of immune checkpoints including programmed cell death protein-1 (PD1), cytotoxic T-lymphocyte-associated protein-4 (CTLA4), T-cell immunoglobulin and mucin-domain containing-3 (TIM3), lymphocyte-activation gene-3 (LAG3), T-cell immunoreceptor with immunoglobulin and ITIM domains (TIGIT), and CD160. This phenomenon was observed in many cancer cells to escape from antitumor immune responses.

The poliovirus receptor (PVR), also known as CD155, is an immunoglobulin -like adhesion molecule, with an important regulatory role in T-cell and natural killer (NK) cell functions, cell migration and proliferation. It is a major ligand that is expressed on epithelial and myeloid cells of the tumor. PVR is able to bind CD226, DNAX accessory molecule-1 (DNAM-1), T-cell-Activated Increased Late Expression Protein (TACTILE), and TIGIT. Binding to DNAM-1 induces the release of pro-inflammatory cytokines and cytotoxicity of T-cells and NK cells (T-cell activation), while binding to TIGIT induces a rather anti-inflammatory, non-proliferative, and noncytotoxic profile (T-cell exhaustion).

CD155 expression was associated with an unfavorable prognosis in solid tumors such as colon cancer, breast cancer, lung adenocarcinoma, pancreatic cancer, melanoma, and glioblastoma, as it correlated with tumor migration, development of metastases, tissue and lymph node invasion, relapse, and poorer survival.

Stamm et al., demonstrated that high CD155 (PVR) expression correlated with poor outcome in AML. Stamm et al., also showed that antibody blockade of PVR on AML cell lines or primary AML cells or TIGIT blockade on immune cells increased the anti-leukemic effects mediated by purified CD3+ cells in vitro. Zhang et al., assessed the prognostic significance and immune-associated mechanism of CD155 and identified that CD155 was commonly upregulated in most human cancers including AML, and high expression of CD155 was closely correlated with unfavorable clinical outcomes.

Our aim is to study the prognostic and predictive values of CD155 expression in AML patients in our locality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed AML.
* Age group: patients more than 18 years old and less than 60 years.
* Patients receiving induction chemotherapy 3&7 at South Egypt Cancer Institute.

Exclusion Criteria:

* Patients less than 18 years old and over 60 years.
* Patients with concurrent malignancy.
* Secondary AML.
* Acute Promyelocytic leukemia (AML-M3).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients (18 - 60 years old) diagnosed as AML
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
CD155 expression in AML | 2 years
  Study the CD155 expression by flow cytometry

SECONDARY OUTCOMES:
CD155 expression with patients' clinical data | 2 years
  Correlation of CD155 expression with clinical, hematological and cytogenetic data of AML patients
CD155 expression and survival | 2 years
  Correlation of CD155 expression levels with patients' outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nehal Rayan, M.D., Principal Investigator — Assistant Lecturer
Locations (1):
- South Egypt Cancer Institute, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dougall WC, Kurtulus S, Smyth MJ, Anderson AC. TIGIT and CD96: new checkpoint receptor targets for cancer immunotherapy. Immunol Rev. 2017 Mar;276(1):112-120. doi: 10.1111/imr.12518. PMID 28258695
- [Background] Gao J, Zheng Q, Xin N, Wang W, Zhao C. CD155, an onco-immunologic molecule in human tumors. Cancer Sci. 2017 Oct;108(10):1934-1938. doi: 10.1111/cas.13324. Epub 2017 Aug 18. PMID 28730595
- [Background] Gorvel L, Olive D. Targeting the "PVR-TIGIT axis" with immune checkpoint therapies. F1000Res. 2020 May 13;9:F1000 Faculty Rev-354. doi: 10.12688/f1000research.22877.1. eCollection 2020. PMID 32489646
- [Background] Li XY, Das I, Lepletier A, Addala V, Bald T, Stannard K, Barkauskas D, Liu J, Aguilera AR, Takeda K, Braun M, Nakamura K, Jacquelin S, Lane SW, Teng MW, Dougall WC, Smyth MJ. CD155 loss enhances tumor suppression via combined host and tumor-intrinsic mechanisms. J Clin Invest. 2018 Jun 1;128(6):2613-2625. doi: 10.1172/JCI98769. Epub 2018 May 14. PMID 29757192 (Retraction: PMID 35289314 J Clin Invest. 2022 Mar 15;132(6):)
- [Background] Liu L, Chang YJ, Xu LP, Zhang XH, Wang Y, Liu KY, Huang XJ. T cell exhaustion characterized by compromised MHC class I and II restricted cytotoxic activity associates with acute B lymphoblastic leukemia relapse after allogeneic hematopoietic stem cell transplantation. Clin Immunol. 2018 May;190:32-40. doi: 10.1016/j.clim.2018.02.009. Epub 2018 Mar 15. PMID 29477343
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Zhang H, Yang Z, Du G, Cao L, Tan B. CD155-Prognostic and Immunotherapeutic Implications Based on Multiple Analyses of Databases Across 33 Human Cancers. Technol Cancer Res Treat. 2021 Jan-Dec;20:1533033820980088. doi: 10.1177/1533033820980088. PMID 33576304
- [Result] Bakhshaei P, Kazemi MH, Golara M, Abdolmaleki S, Khosravi-Eghbal R, Khoshnoodi J, Judaki MA, Salimi V, Douraghi M, Jeddi-Tehrani M, Shokri F. Investigation of the Cellular Immune Response to Recombinant Fragments of Filamentous Hemagglutinin and Pertactin of Bordetella pertussis in BALB/c Mice. J Interferon Cytokine Res. 2018 Apr;38(4):161-170. doi: 10.1089/jir.2017.0060. PMID 29638208